CLINICAL TRIAL: NCT04779580
Title: Optimising Analgesia for Lateral Hip Arthroplasty Incision: Can a Subcostal Nerve Block Add Benefit to a Lateral Femoral Cutaneous Nerve Block?
Brief Title: Can a Subcostal Nerve Block Add Benefit to a Lateral Femoral Cutaneous Nerve Block for Open Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Queen Elizabeth Hospital King's Lynn NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSBF01
Record Dates: First submitted 2021-02-21; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia, Local
Keywords: Regional Anaesthesia; Hip Surgery; Lateral Femoral Cutaneous Nerve; Subcostal Nerve; Analgesia; Hip Arthroplasty
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Only Group) (Experimental): Only one group in this study. 10 participants to have intervention.
  Lateral femoral cutaneous nerve block and evaluation:
  Routine ECG, pulse oximetry and blood pressure monitoring will be available. Using a sterile technique, the lateral femoral nerve will be approached using an in-plane ultrasound-guided technique, using a Stimuplex Ultra 360 50mm needle (B Braun, UK). Following negative aspiration, a one off STAT injection of 5mls lidocaine 1% will be administered subcutaneously.
  After 10 minutes, any altered sensation will be assessed using ice to differentiate normal and altered sensation. This area will be marked on the skin using a black marker pen. Photographs will be taken and images of the procedure will be recorded.
  The above will then be repeated for the subcostal nerve block.
  The total area of anaesthesia will then be compared to the standard surgical incision for hip surgery to assess whether the subcostal nerve block will offer any further analgesia.
  Interventions: Procedure: Lateral Cutaneous Nerve Of The Thigh Nerve Block Using Local Anaesthetic; Procedure: Subcostal Nerve Block Using Local Anaesthetic

INTERVENTIONS:
Procedure: Lateral Cutaneous Nerve Of The Thigh Nerve Block Using Local Anaesthetic — Currently accepted aseptic conditions will be met. The lateral cutaneous nerve of the thigh will be identified on ultrasound (Sonosite X-Porte) and 5mL of 1% lidocaine will be administered around the nerve using a 50mm Stimuplex needle. The area of anaesthesia will be demarcated using ice.
Procedure: Subcostal Nerve Block Using Local Anaesthetic — Currently accepted aseptic conditions will be met. The subcostal nerve will be identified on ultrasound (Sonosite X-Porte) and 5mL of 1% lidocaine will be administered around the nerve using a 50mm Stimuplex needle. The area of anaesthesia will be demarcated using ice.

SUMMARY:
Hip Surgery is a very common form of surgery carried out across many hospitals within the UK in emergency and elective form. There is a variation between amongst surgeons with regard to the initial surgical incision required for the operation. It is fairly common practice to anaesthetise the Lateral Cutaneous Nerve of the thigh for analgesic reasons prior to the start of surgery, however due to the variation in surgical practice (and evolving surgical practices) this may not cover the entire surgical incision site. Another group of nerves termed the subcostal nerves has been described in the texts to perhaps cover the area of surgical incision along with blockade of the lateral cutaneous nerve of the thigh. On healthy volunteers the investigators plan to anaesthetise the lateral cutaneous nerve of the thigh, and the subcostal nerve on healthy participants to ascertain and map out the area of anaesthesia to see whether this could be a viable technique for analgesia for hip surgery in the future.

DETAILED DESCRIPTION:
Hip replacement and hemiarthroplasty of the hip for neck of femur fracture are common orthopaedic procedures. The National Joint Registry in 2017 reported that 96.3% of hip replacements were performed using the anterolateral and posterior approach. NICE guidelines have suggested to utilise the anterolateral approach for hip fracture hemiarthroplasty due to decrease dislocation rates and thus, cost savings.

Despite these two commonly use approaches, the traditional incisions have, in the investigators experience, been modified. This is to accommodate the increasing evidence and emphasis on the acetabular components. Besides that, in hemiarthroplasty, various incisions have been described for the 'anterolateral' approach, such as direct lateral, curved posteriorly. 'Mini' and 'micro' incisions of the posterior approach has also been described all with the aim as tissue-sparing procedures, improving outcomes and length of stay.

In this study, the investigators aim to describe the 'traditionally' described posterior and anterolateral incisions to the hip by Moore and Hardinge:

1. Posterior - 5cm distally from the greater trochanter along the femoral diaphysis, curving the incision proximally 3-8cm towards the PSIS
2. Anterolateral - 3cm distally from the greater trochanter along the femoral diaphysis, continuing proximally 3-8cm along the femoral diaphysis

The cutaneous innervation for this area is largely supplied by the lateral femoral cutaneous nerve of the thigh; however some anatomical texts also describe contribution to this area from the subcostal nerve, or the lateral branches of the iliohypogastric nerve.

The lateral femoral cutaneous nerve can be readily identified using ultrasound, and has recently been categorised into 3 distinct types; the 'Sartorius', Posterior' and the 'Fan' types. The Sartorius type, accounting for roughly one-third, describes a dominant anterior branch running along the border of the Sartorius muscle, with no or few posterior branches.

The posterior type, accounting for roughly one-third, describes a strong posterior branch, equal in thickness to, or thicker than, the anterior branch running laterally and crossing the medial border of the tensor fasciae latae muscle immediately distal to the ASIS.

The fan type, accounting for roughly one-third, describes multiple nerve branches of equal thickness spreading over the anterolateral region of the proximal aspect of the thigh, crossing over the tensor fasciae latae muscle and the lateral border of the sartorius.

The lateral femoral cutaneous nerve can readily be identified using ultrasound and is readily blocked.

The subcostal nerve describes the distal continuation of the twelfth intercostal nerve.

Its lateral cutaneous branch perforates the obliquus internus and externus, descends over the iliac crest in front of the lateral cutaneous branch of the iliohypogastric, and is distributed to the skin of the front part of the gluteal region, extending as low as the greater trochanter.

The iliohypogastric nerve is usually a branch of the lumbar plexus originating from the L1 ventral ramus. Above the iliac crest, it enters the posterior part of the transversus abdominis. Between the transversus abdominis and internal oblique it divides into lateral and anterior cutaneous branches. The lateral cutaneous branch runs through the internal and external oblique above the iliac crest, a little behind the iliac branch of the T12 spinal nerve. It is distributed to the posterolateral gluteal skin. The iliohypogastric nerve usually gives communicating branches to the subcostal and ilioinguinal nerves. The iliac branch of the iliohypogastric nerve can be absent, replaced by the lateral cutaneous branch of the subcostal nerve. The iliohypogastric nerve is sometimes derived from the twelfth thoracic nerve and can also receive a root from the eleventh. Anloague and Huijbregts (2009) demonstrated the absence of the iliohypogastric nerve in 20.6% of the lumbar plexuses they investigated.

Anaesthesia for this incision can therefore only partly be achieved by a lateral femoral cutaneous nerve block; however this is not always complete for the territory of the incision, particularly if the incision is longer and extending more proximally. Due to the variation and sharing between the subcostal and iliohypogastric nerves, and their similar course, we will consider sonographically identified descending nerves to the gluteal region as a single entity, referred to as the subcostal nerve.

The Investigators have identified the subcostal nerve using ultrasound on volunteers and found it to lie above the superficial fascia directly above gluteus medius at the cranial aspect of the buttock, originating from the lateral abdominal wall musculature, where it can be tracked proximally to visualise its descent through the muscle layers of the lateral abdominal wall.

The investigators hypothesise that a lateral femoral cutaneous nerve block alone will not reliably provide cutaneous anaesthesia to the territory of our commonly observed incisions for hip arthroplasty. Our secondary hypothesis is that a blockade of the subcostal nerve will extend the cutaneous anaesthesia to reliably cover that area.

This study is to be conducted in three parts. Firstly, surgeons within the investigators department will be canvassed to mark out their likely line of incision for a routine elective primary hip arthroplasty. Pictorial evidence and variation will be gathered for overlay. Secondly, on volunteers, the lateral femoral cutaneous nerve will be identified using ultrasound in its course distal to the inguinal ligament, and the relevant type will be ascertained. The nerve will then be blocked using a short-acting local anaesthetic, and the area of numbness demarcated. Pictorial evidence will be gathered.

Thirdly, the subcostal nerve will be identified, and blocked using a short-acting local anaesthetic. The resulting area of numbness will be further demarcated, and further pictorial evidence gathered.

The relevant demarcated areas and incisions will be then be compared for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Peripheral neuropathy of any aetiology
* Diabetes mellitus
* Meralgia paraesthetica
* Previous Total Hip Arthroplasty
* Sciatica
* Spinal Stenosis
* Localised infection of the inguinal or gluteal regions
* Allergy to local anaesthetic or excipients
* Inability to identify either the lateral femoral cutaneous nerve or the subcostal nerve using ultrasound

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Cutaneous area anaesthetised by lateral cutaneous nerve of thigh and subcostal nerve block using local anaesthetic | Duration of Study (approximately 5 months)
  Demarcated area of sensory loss after lateral femoral cutaneous nerve block and subcostal nerve block - reported by the participant upon testing the area with cold ice by the investigators. The area will then be assessed by the investigators to assess whether the area of anaesthesia will cover the surgical incision site for hip arthroplasties.

CONTACTS AND LOCATIONS:
Overall Officials: James Stimpson, FRCA, Principal Investigator — Queen Elizabeth Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Rudin D, Manestar M, Ullrich O, Erhardt J, Grob K. The Anatomical Course of the Lateral Femoral Cutaneous Nerve with Special Attention to the Anterior Approach to the Hip Joint. J Bone Joint Surg Am. 2016 Apr 6;98(7):561-7. doi: 10.2106/JBJS.15.01022. PMID 27053584
- [Background] Ray B, D'Souza AS, Kumar B, Marx C, Ghosh B, Gupta NK, Marx A. Variations in the course and microanatomical study of the lateral femoral cutaneous nerve and its clinical importance. Clin Anat. 2010 Nov;23(8):978-84. doi: 10.1002/ca.21043. PMID 20830791
- [Background] Bodner G, Bernathova M, Galiano K, Putz D, Martinoli C, Felfernig M. Ultrasound of the lateral femoral cutaneous nerve: normal findings in a cadaver and in volunteers. Reg Anesth Pain Med. 2009 May-Jun;34(3):265-8. doi: 10.1097/AAP.0b013e31819a4fc6. PMID 19587628
- [Background] Anloague PA, Huijbregts P. Anatomical variations of the lumbar plexus: a descriptive anatomy study with proposed clinical implications. J Man Manip Ther. 2009;17(4):e107-14. doi: 10.1179/106698109791352201. PMID 20140146